CLINICAL TRIAL: NCT06249724
Title: Noninvasive Modulation of Chronic Neuropathic Pain With Focused Ultrasonic Waves
Brief Title: Noninvasive Modulation of Chronic Neuropathic Pain
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Not activated at the site level
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jan Kubanek, Assistant Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00175546
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Neuropathic Pain; Chronic Pain
MeSH Terms: conditions — Neuralgia; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active stimulation (Active Comparator): Low-intensity focused ultrasound stimulation of dorsal root ganglion involved in pain conduction
  Interventions: Device: Active stimulation using low-frequency ultrasonic transducer
- Sham stimulation (Sham Comparator): Zero-intensity focused ultrasound stimulation of dorsal root ganglion involved in pain conduction
  Interventions: Device: Sham stimulation using low-frequency ultrasonic transducer

INTERVENTIONS:
Device: Active stimulation using low-frequency ultrasonic transducer — The ultrasonic transducer delivers focused low-intensity ultrasound stimulation
  Arms: Active stimulation
Device: Sham stimulation using low-frequency ultrasonic transducer — The ultrasonic transducer delivers focused zero-intensity ultrasound stimulation
  Arms: Sham stimulation

SUMMARY:
This study will apply low-intensity transcranial focused ultrasound to dorsal root ganglia in patients with chronic neuropathic pain. The target will be validated using magnetic resonance imaging. The stimulation will first be delivered using a range of stimulation parameters during psychophysical and physiological monitoring. A well-tolerated stimulation protocol will be selected for subsequent testing in a blinded randomized sham-controlled cross-over trial. The level of pain will be evaluated using the Numerical Rating Scale (NSR-11) and the Patient-Reported Outcomes Measurement Information System (PROMIS) numerical rating scales of pain.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of chronic pain
* Moderate-to-severe chronic pain lasting at least 2 months
* Stated willingness to comply with all study procedures and avoid changes to current treatments (medications, physical therapy, cognitive behavioral therapy) for the duration of the study
* For females of reproductive potential: negative pregnancy test or use of highly effective contraception for at least 1 month prior to baseline; agreement to use such a method throughout the study
* Capacity to provide informed consent; provision of a signed and dated consent form

Exclusion Criteria:

* Poorly managed general medical condition
* Pregnant or breast feeding
* Implanted device in the back
* Lifetime history of a serious suicide attempt
* Clinically inappropriate for participation in the study as determined by the study team

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity: momentary change | During the intervention, and every day thereafter, for 7 days
  Numerical Rating Scale (NRS-11) of pain. NRS-11 is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Pain intensity: subjective state | Immediately after the intervention, and every day thereafter, for 7 days
  PROMIS scale of pain intensity. Scores range from 1 (no pain) to 5 (severe pain). A lower score indicates a better treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kubanek, PhD, Principal Investigator — University of Utah; Daniel Odell, MD, Study Chair — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No